CLINICAL TRIAL: NCT06202729
Title: Focus on Experienced Anxiety Related to an Emergency Department Visit
Acronym: FEAR-ED
Status: Completed | Type: Observational
Sponsor: Frisius Medisch Centrum (Other)
Responsible Party: Sponsor
Other Study IDs: MCLSEH1
Record Dates: First submitted 2023-12-15; First posted 2024-01-11 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Fear
Keywords: Fear, anxiety
MeSH Terms: conditions — Anxiety Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — GAD-7, VAS-A, NRS

SUMMARY:
The aim of the present study is to determine the prevalence of anxiety in adult patients attending the ED of the Medical Centre Leeuwarden.

DETAILED DESCRIPTION:
Determination of the prevalence of anxiety in adult patients attending the ED of the Medical Centre Leeuwarden. Secondarily, the common causes of anxiety and the effect of anxiety on the time of presentation to the ED and perceived pain will be investigated. In addition to gaining more insight into the relationship between the ED and anxiety, the study aims to raise awareness of anxiety among patients in the ED.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Competent to decide on study participation
* Written informed consent obtained

Exclusion Criteria:

* Patients from who a Dutch questionnaire cannot be obtained (e.g. delirious, comatose, confused and non-Dutch speaking patients)
* If the reason for ED presentation is: suicide, intoxication or reporting from a sexual violence center
* Patients with an active eating disorder
* Patient already included in this study
* Objection to the use of patient data registered in the EPD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients visiting the ED.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2023-12-11 (Actual)

PRIMARY OUTCOMES:
Prevalence of anxiety measured by GAD-7 and VAS-A | Two weeks prior to ED presentation
  What is the prevalence of anxiety among adult patients in the ED?

SECONDARY OUTCOMES:
Timing ER visit | 1 Day
  What influence does fear have on the timing of the ER visit?
Start of fear (open question) | 1 Day
  What was the moment when fear arised?
Influence of pain (NRS) on fear (GAD-7) | 1 Day
  What is the influence of pain on fear experienced?
Cause of fear (open question) | 1 Day
  What is the cause of fear?

CONTACTS AND LOCATIONS:
Locations (1):
- MCLeeuwarden, Leeuwarden, Provincie Friesland, Netherlands

IPD SHARING:
Plan to Share IPD: No